CLINICAL TRIAL: NCT01782391
Title: Impact of Transcranial Slow Oscillating Stimulation on Memory Consolidation During Nocturnal Slow Wave Sleep in Patients With Mild Cognitive Impairments(MCI)
Brief Title: Effects of Brain Stimulation During Nocturnal Sleep on Memory Consolidation in Patients With Mild Cognitive Impairments
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of appropriate participants
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Agnes Flöel, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Nighttime sleep-tSOS-MCI
Record Dates: First submitted 2012-06-05; First posted 2013-02-01 (Estimated); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Mild Cognitive Impairment, So Stated
Keywords: mild cognitive impairment; dementia; MCI; brain stimulation; tSOS; tDCS; sleep; memory; memory consolidation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0,75 Hz stimulation (Experimental): slow transcranial oscillating stimulation (~0,75Hz) during periods of Slow Wave Sleep
  Interventions: Device: Stimulation
- SHAM stimulation (Sham Comparator): SHAM stimulation during periods of Slow Wave Sleep
  Interventions: Device: SHAM

INTERVENTIONS:
Device: Stimulation
  Other Names: oscillating direct current brain stimulation
  Arms: 0,75 Hz stimulation
Device: SHAM — no stimulation
  Arms: SHAM stimulation

SUMMARY:
The beneficial effect of nocturnal sleep on memory consolidation is well-documented in young, healthy subjects. Especially, periods rich in slow-wave sleep (SWS) have shown a memory enhancing effect on hippocampus-dependent declarative memory. Slow oscillatory activity typically occuring during SWS has been implicated in the consolidation effect. Recent evidence in young healthy subjects suggest that the sleep-associated consolidation effect can be amplified by the application of a weak transcranial oscillatory electric current within the frequency range of SWS in humans (0,7-0,8 Hz) during SWS. If patients with amnestic mild cognitive impairments (MCI)- usually characterized by initial difficulties in hippocampus dependent memory functions - benefit from transcranial slow oscillatory stimulation (tSOS) during nocturnal sleep as well has not been studied so far. The primary aim of the present study is to investigate the influence of a weak slow oscillating brain stimulation (tSOS) on declarative memory consolidation applied during periods of nocturnal SWS in MCI patients.

ELIGIBILITY:
Inclusion Criteria:

* amnestic and amnestic plus MCI-patients:

  1. Concern reflecting a change in cognition reported by patient or informant or clinician (i.e., historical or observed evidence of decline over time)
  2. Objective evidence of memory impairment; additional cognitive domains may be affected as well;
  3. Preservation of independence in functional abilities
  4. no dementia
* age: 50-90 years

Exclusion Criteria:

* untreated severe internal or psychiatric diseases
* epilepsy
* other severe neurological diseases eg., previous major stroke, brain tumour
* dementia
* contraindications to MRI

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Retention of declarative memories after 0.75 Hz stimulation during SWS, vs after sham stimulation during SWS | 4 weeks
  Retention between stimulation conditions (0.75 Hz during SWS, vs sham stimulation during SWS) in the declarative memory task.

SECONDARY OUTCOMES:
Amount of Slow wave Sleep, spindels, eeg-correlates, further memory systems | 4 weeks
  1. Amount of slow wave sleep assessed by standard polysomnographic criteria in 0,75 Hz vs SHAM stimulation during SWS.
  2. Spindel activity during sleep indicated via several spindel parameters like number, duration, frequency of spindles; compared between 0,75 Hz and SHAM stimulation during SWS.
  3. Neuronal correlates (EEG-power in slow oscillation frequency bands induced by 0,75 Hz vs SHAM stimulation during SWS; EEG-correlates of encoding and retrieval of a declarative memory task).
  4. Performance in further memory systems (procedural), compared between 0,75 Hz and SHAM stimulation during SWS.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Professor, Study Chair — Charite Universitätsmedizin Berlin - Neurologie
Locations (1):
- Charite CCM Neurologie Berlin, Berlin, Germany

REFERENCES:
- [Background] Boggio PS, Khoury LP, Martins DC, Martins OE, de Macedo EC, Fregni F. Temporal cortex direct current stimulation enhances performance on a visual recognition memory task in Alzheimer disease. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):444-7. doi: 10.1136/jnnp.2007.141853. Epub 2008 Oct 31. PMID 18977813
- [Background] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Background] Naismith SL, Lewis SJ, Rogers NL. Sleep-wake changes and cognition in neurodegenerative disease. Prog Brain Res. 2011;190:21-52. doi: 10.1016/B978-0-444-53817-8.00002-5. PMID 21531243